CLINICAL TRIAL: NCT06654882
Title: Trial of Sequential Medications AfteR TNFi Failure in Juvenile Idiopathic Arthritis
Acronym: SMART-JIA
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Pro00115808; PLACER-2022C3-30331 (Other Grant/Funding Number: PCORI); EPM #8533 (Other Grant/Funding Number: DukeUMC)
Record Dates: First submitted 2024-10-21; First posted 2024-10-23 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2024-10

CONDITIONS: Polyarticular Course Juvenile Idiopathic Arthritis (JIA)
Keywords: JIA; Rheumatology
MeSH Terms: conditions — Arthritis, Juvenile | interventions — Tumor Necrosis Factor Inhibitors; Dosage Forms; Abatacept; tocilizumab; tofacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Second TNFi (Tumor Necrosis Factor inhibitor) medication (Active Comparator): Adalimumab originator or biosimilar; etanercept originator or biosimilar depending on which TNFi the participant had failed.
  Interventions: Drug: TNFi (Tumor Necrosis Factor inhibitor) medication
- Abatacept (Active Comparator): The 50 mg, 87.5 mg and 125 mg SQ doses will be available for weight-based dosing. All participants randomized to abatacept in the first or second stage randomization will receive abatacept SQ weekly at a dosage based on the participant's body weight
  Interventions: Drug: Abatacept
- Tocilizumab originator or biosimilar (Active Comparator): Tocilizumab will be provided in prefilled syringes (162 mg tocilizumab/0.9 mL solution). All participants randomized to tocilizumab in the first or second stage randomization will be receiving 1 prefilled syringe (162 mg) with a dosing interval based on the body weight criteria.
  Interventions: Drug: Tocilizumab
- Tofacitinib (Active Comparator): Tofacitinib will be provided as oral tablets (tofacitinib citrate 5 mg) and as an oral solution (1 mg/mL). All participants randomized to tofacitinib in the first or second stage randomization will receive tofacitinib oral tablets or oral solution twice daily, approximately 12 hours apart, in the morning and evening, at a dosage based on the participant's body weight .
  Interventions: Drug: Tofacitinib

INTERVENTIONS:
Drug: TNFi (Tumor Necrosis Factor inhibitor) medication — Adalimumab 10 kg (22 lbs) to <15 kg (33 lbs) 10 mg every other week* 15 kg (33 lbs) to <30 kg (66 lbs) 20 mg every other week ≥30 kg (66 lbs) 40 mg every other week
  Etanercept
  ≥63 kg (138 lb) 50 mg weekly <63 kg (138 lb) 0.8 mg/kg weekly
  Arms: Second TNFi (Tumor Necrosis Factor inhibitor) medication
Drug: Abatacept — 10 kg to <25 kg 50 mg once weekly 25 kg to <50 kg 87.5 mg once weekly
  ≥50 kg 125 mg once weekly
  Arms: Abatacept
Drug: Tocilizumab — <30 kg 162 mg once every 3 weeks
  ≥30 kg 162 mg once every 2 weeks
  Arms: Tocilizumab originator or biosimilar
Drug: Tofacitinib — 10 to <20 kg 3.2 mg (3.2 mL oral solution) BID 20 to <40 kg 4 mg (4 mL oral solution) BID
  ≥40 kg 5 mg (one 5 mg tablet or 5 mL oral solution) BID
  Arms: Tofacitinib

SUMMARY:
This study is an open-label, randomized, multicenter trial that incorporates a multi-arm design comparing each of 3 non-TNFi (Tumor Necrosis Factor inhibitor) medications to a second TNFi (active control) within a sequential multiple assignment randomized trial design with 2 randomization stages corresponding with clinical decision points. The first randomization addresses whether each of the 3 non-TNFi medications is superior to treatment with a second TNFi. The second randomization allows identification of optimal sequential use of biologics (treatment strategies).

DETAILED DESCRIPTION:
The goal of the study is to provide an evidence base for selecting sequential medication(s) if a JIA patient fails initial bDMARD. SMART-JIA is a pragmatic, international, open-label, randomized trial comparing treatment with a second TNFi (active control) to each of 3 different medications (IL-6i, JAKi, or ABA) in children aged 2 to 17 years with pcJIA and inadequate response to initial TNFi. Leveraging sequential multiple assignment randomized trial (SMART) design methodology, we will implement a second randomization to assess the effectiveness of changing medication if there is inadequate response to the first study medication. This approach allows identification of optimal strategies for medication sequencing based on individual characteristics and provides critical insights to inform future studies.

SMART-JIA will study the efficacy of a second TNFi (active control) compared to each of 3 other already US Food and Drug Administration (FDA)-approved and European Union (EU)-approved non-TNFi medications currently used to treat pcJIA (IL-6i, JAKi, and ABA). TNFi, IL-6i, and ABA are administered by subcutaneous (SQ) injection weekly, or every other week, or every three weeks, and JAKi (e.g., tofacitinib) is taken orally twice daily. All study treatments have similar safety profiles and are standard of care (SOC) worldwide. This in addition to the pragmatic and full-scale nature of the trial will ensure its completion. Successful completion of this trial will substantially impact the clinical care and outcomes of children with pcJIA, shifting the current trial-and-error treatment paradigm to a smart, precise approach.

ELIGIBILITY:
Inclusion Criteria:

* Polyarticular course JIA
* Moderate or high-disease activity (cJADAS10 >5) despite treatment with an initial TNFi for ≥3 months
* Age ≥2 years and <18 years and weight ≥ 10kg
* No systemic glucocorticoids or systemic glucocorticoids at a stable dose of ≤0.2 mg/kg/day (maximum 10 mg/day) for ≥2 weeks prior to baseline visit
* Documented informed consent/assent obtained from the parent/caregiver/patient

Exclusion Criteria:

* Systemic JIA
* Enthesitis-related arthritis/juvenile spondyloarthritis (2001 International League of Associations for Rheumatology [ILAR] criteria)30
* History of or currently active inflammatory bowel disease
* History of or currently active psoriasis
* Active uveitis within 3 months of the baseline visit
* History of or currently active sacroiliitis
* History of or current malignancy
* Active tuberculosis (TB) or a history of incompletely treated TB; Purified Protein derivative (PPD) or QuantiFERON-TB positive patients (without active TB) unless it is documented that the patient has been adequately treated for TB and can start treatment with a biologic agent, based on the medical judgment of the site investigator and/or an infectious disease specialist; suspected extrapulmonary TB infection; or at high risk of contracting TB, such as close contact with individual with active or latent TB
* Prior treatment with more than one TNFi molecule; exposure to more than one biosimilar of the same TNFi molecule is allowed
* Prior treatment with non-TNFi bDMARDs and/or any JAKi
* Aspartate aminotransferase (AST) or alanine transaminase (ALT) ≥3 × upper limit of normal (ULN) for age and sex
* Serum creatinine >1.5 × ULN for age and sex
* Platelet count <150 × 103/μL (<150,000/mm3)
* Hemoglobin <7.0 g/dL (<4.3 mmol/L)
* White blood cell (WBC) count <3,000/mm3 (<3.0 × 109/L)
* Neutrophil count <1,500/mm3 (<1.5 × 109/L)
* Any active acute, subacute, chronic, or recurrent bacterial, viral, or systemic fungal infection or any major episode of infection requiring hospitalization or treatment during screening or treatment with IV antibiotics completed within 4 weeks of the screening visit or oral antibiotics completed within 2 weeks of the screening visit
* Any medical history that may be considered a contraindication/safety concern with the use of adalimumab, etanercept, tofacitinib, ABA, or an IL-6 inhibitor or their biosimilars, in the opinion of the site investigator

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 400 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with MiDA | Month 6
  Minimal disease activity (MiDA) at Month 6 as assessed by the cJADAS10 ≤5
  MiDA is low-disease activity and inactive disease in this protocol.
  Score range for the cJADAS10 (total): 0 - 30.
  Disease State cJADAS10 Score Inactive disease ≤2.5 Low-disease activity 2.6 - 5 Moderate-disease activity 5.1 - 16 High-disease activity >16
  Minimal disease activity (MiDA) is a state of low disease activity or remission that is considered a useful treatment target for both patients and physicians.
  The clinical Juvenile Arthritis Disease Activity Score (cJADAS10) is a tool used to measure the level of disease activity in non-systemic juvenile idiopathic arthritis (JIA). It's a composite index that combines information from several sources, including:
  * The number of active joints, up to 10
  * The physician's global assessment of disease activity (PhGA)
  * The patient or parental global assessment of well-being (PaGA)

SECONDARY OUTCOMES:
PROMIS® Pain Interference at Month 6 | Month 6
  Patient-Reported Outcomes Measurement Information System (PROMIS).
  For most PROMIS instruments, a score of 50 is the average for the United States general population with a standard deviation of 10 because calibration testing was performed on a large sample of the general population.
  For PROMIS measures, higher scores equals more of the concept being measured (e.g., more Fatigue, more Physical Function). Thus a score of 60 is one standard deviation above the average referenced population. This could be a desirable or undesirable outcome, depending upon the concept being measured.
PROMIS® Fatigue at Month 6 | Month 6
  Patient-Reported Outcomes Measurement Information System (PROMIS).
  For most PROMIS instruments, a score of 50 is the average for the United States general population with a standard deviation of 10 because calibration testing was performed on a large sample of the general population.
  For PROMIS measures, higher scores equals more of the concept being measured (e.g., more Fatigue, more Physical Function). Thus a score of 60 is one standard deviation above the average referenced population. This could be a desirable or undesirable outcome, depending upon the concept being measured.
PROMIS® Physical Function at Month 6 | Month 6
  Patient-Reported Outcomes Measurement Information System (PROMIS).
  For most PROMIS instruments, a score of 50 is the average for the United States general population with a standard deviation of 10 because calibration testing was performed on a large sample of the general population.
  For PROMIS measures, higher scores equals more of the concept being measured (e.g., more Fatigue, more Physical Function). Thus a score of 60 is one standard deviation above the average referenced population. This could be a desirable or undesirable outcome, depending upon the concept being measured.
Change in arthritis disease activity (cJADAS10) | Month 6
  Minimal disease activity (MiDA) at Month 6 as assessed by the cJADAS10 ≤5
  MiDA is low-disease activity and inactive disease in this protocol.
  Score range for the cJADAS10 (total): 0 - 30.
  Disease State cJADAS10 Score Inactive disease ≤2.5 Low-disease activity 2.6 - 5 Moderate-disease activity 5.1 - 16 High-disease activity >16
  Minimal disease activity (MiDA) is a state of low disease activity or remission that is considered a useful treatment target for both patients and physicians.
Change in arthritis disease activity (JIA American College of Rheumatology Pediatric 70 [ACR 70]) at Month 6 | Month 6
  The ACR score is a scale to measure change in rheumatoid arthritis symptoms.
  An ACR70 response represents at least a 70% improvement in tender and swollen joint counts.
Number of participants with MiDA (Change in arthritis disease activity [cJADAS10] at Month 12) | Month 12
  Minimal disease activity (MiDA) at Month 12 as assessed by the cJADAS10 ≤5
  MiDA is low-disease activity and inactive disease in this protocol.
  Score range for the cJADAS10 (total): 0 - 30.
  Disease State cJADAS10 Score Inactive disease ≤2.5 Low-disease activity 2.6 - 5 Moderate-disease activity 5.1 - 16 High-disease activity >16
  Minimal disease activity (MiDA) is a state of low disease activity or remission that is considered a useful treatment target for both patients and physicians.

IPD SHARING:
Plan to Share IPD: No